CLINICAL TRIAL: NCT02445950
Title: With-Me - Technology-Aided Phone Coaching for Occupational Health Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VTT Technical Research Centre of Finland (Other)
Collaborators: Firstbeat Technologies Ltd. (Industry); Mawell Care Ltd (Unknown); Mawell Ltd (Unknown); Oulun Työterveys (Unknown); Technical University of Denmark (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 332885 With-Me-Occ
Record Dates: First submitted 2015-05-06; First posted 2015-05-15 (Estimated); Last update posted 2016-04-26 (Estimated); Status verified 2016-04

CONDITIONS: Psychological Stress
Keywords: Coaching; Well-being; Digital Health; Profiling; Customer Satisfaction; User Experience; Occupational Health; Lifestyle; Psychological Stress; Cost-Effectiveness; Guideline Adherence
MeSH Terms: conditions — Stress, Psychological; Consumer Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Technology-aided counseling (Experimental): Customers receive intervention via technology-aided phone wellness counseling. The intensive phase lasts 13 weeks and includes 5 phone calls. The customers are able to view their change change needs and choose tasks/goals for the coaching. The independent phase lasts 13 weeks and coaching is done via a digital tool.
  Interventions: Behavioral: Technology-aided phone wellness counselling
- Traditional counseling (Active Comparator): Customers receive intervention via traditional phone wellness counseling. The intensive phase lasts 13 weeks and includes 5 phone calls. Change needs and goals are set during the phone calls. The independent phase lasts 13 weeks and includes 3 phone calls.
  Interventions: Behavioral: Phone wellness counselling

INTERVENTIONS:
Behavioral: Technology-aided phone wellness counselling — The intervention provides phone wellness counselling with the help of web-based interventions, digital profiling and suggestion tool in occupational health.
  Arms: Technology-aided counseling
Behavioral: Phone wellness counselling — The intervention provides phone wellness counseling in occupational health.
  Arms: Traditional counseling

SUMMARY:
The purpose of this study is to examine whether the technology (web-based coaching, profiling and suggestion tool) brings added value to the traditional phone coaching in occupational health context. The interventions are phone counseling interventions. The other intervention exploits additionally a specific web-based coaching, profiling and suggestion tool.

DETAILED DESCRIPTION:
The study focuses on mental well-being. The both interventions include intensive and independent phase.

The intensive phase lasts 13 weeks. In the intensive phase, goals for the coaching are defined. Coach calls the customer every two weeks and they discuss about the actions that took place in the previous two weeks and what they need to do in the next two weeks. In the technology-aided arm, customers get and analysis of their change needs via digital tool. Based on the change needs they receive task/goal suggestions from which they need to choose 3. Coach is able to see these choices and exploits it in the coaching. The selected behavioral activation interventions are delivered to customer utilizing a web-based coaching tool.

The independent phase lasts 13 weeks. In the independent phase, technology-aided group is coached via the digital tool. The phone counseling group gets 3 phone calls.

ELIGIBILITY:
Inclusion Criteria:

* At least a bachelor level degree
* Age over 18 years
* Decreased psycho-physic state (own assessment)
* Is in a relationship
* Motivated to enhance own well-being and willing to change lifestyle, to do exercises related on mental well-being and relationship
* Willing to use technological wellness coaching tools, familiarity with technology

Exclusion Criteria:

* Work includes night shifts
* Acute health conditions or serious diseases
* Chronical pain affecting functionality
* Long period(s) of absence from work during the coaching period (e.g. long vacation, alternation leave, parental leave, pension)
* Participation in some other study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2014-11; Primary Completion 2015-11 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Time used for coaching | 6 months
  Measured by the coaches' working time dedicated to coaching from manual logs and Movendos log. This is used to evaluate the cost of coaching.
Psychological wellbeing | 6 months
  Measured by the Työoptimi occupational health questionnaire. This is used to evaluate the effectiveness of the coaching.

SECONDARY OUTCOMES:
Customer satisfaction for coaching | 6 months
  Measured by ad hoc questionnaires.
Occupational health | 6 months
  Measured by Työoptimi occupational health questionnaire.
Satisfaction to life situation | 6 months
  Measured by scale from 1 to 5.
Self-esteem | 6 months
  Measured by 10-item Rosenberg's Self-Esteem Scale.
Cognitive fusion | 6 months
  Measured by 7-item Cognitive Fusion Questionnaire
Perceived stress | 6 months
  Measured by a single-item stress scale.
Satisfaction to a relationship | 6 months
  The scale is modified from The Family Federation of Finland's quality test of a relationship.
Activeness in conducting tasks | 6 months
  Self-assessment measured via phone interviews and questionnaires.
Carefulness in conducting tasks | 6 months
  Self-assessment measured via phone interviews and questionnaires.
Readiness to change | 6 months
  Readiness to change scale measured by questionnaire based on Transtheoretical Model (Stages of Change).
Lifestyle | 6 months
  Evaluated by ad hoc questionnaire on amount of sleep, alcohol consumption and smoking, and eating habits.
Number of the changes made to the profile | 1 month
  Data from the profiling database.
Perceived Accuracy of the profiling tool | 1 month
  Assessed by the coaches via questionnaires.
Perceived ease of use | 6 months
  Measured by questionnaires to customers, questionnaires and interview to coaches.
Perceived usefulness | 6 months
  Measured by the questionnaires to customers, questionnaires and interview to coaches.

CONTACTS AND LOCATIONS:
Overall Officials: Hannu Nieminen, PhD, Principal Investigator — Technical University of Denmark; Jouni Kaartinen, DSc, Principal Investigator — VTT Technical Research Centre of Finland Ltd

REFERENCES:
- [Derived] Muuraiskangas ST, Honka AM, Junno UM, Nieminen HO, Kaartinen JK. A Technology-Assisted Telephone Intervention for Work-Related Stress Management: Pilot Randomized Controlled Trial. J Med Internet Res. 2022 Jul 13;24(7):e26569. doi: 10.2196/26569. PMID 35830233
- See also: Project website — http://www.with-me-project.eu/